CLINICAL TRIAL: NCT06356142
Title: The Effects of Palmar Cooling on Repeated Sprinting Ability
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Jacob B. Daniels DPT, EdD, Assistant Professor, University of Mississippi Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UMMC-IRB-2023-317
Record Dates: First submitted 2024-03-27; First posted 2024-04-10 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2024-06

CONDITIONS: Exercise Induced Fatigue

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Device: Palmar Cooling
- Control (Placebo Comparator)
  Interventions: Device: Placebo Palmar Cooling

INTERVENTIONS:
Device: Palmar Cooling — Palmar cooling device will be utilized for 2 minutes during rest breaks.
  Arms: Intervention Group
Device: Placebo Palmar Cooling — Placebo Palmar cooling device will be utilized for 2 minutes during rest breaks
  Arms: Control

SUMMARY:
Repeated sprinting ability is key for athletic performance in a variety of sport settings. Significant degradations in work output (i.e. fatigue) have been shown to develop after just one sprinting bout1. This pilot study aims to investigate the effects that noninvasive transient temperature manipulation has on an individual's ability to perform repeated sprints. The investigators aim to enroll 90 healthy individuals, 18-30 years of age. Participants will be randomized into two groups (Group A, and B). All groups will perform a ten-minute warm-up followed by two minutes of rest. Following the warm-up and rest period, all groups will participate in a series of five sprints, 60 meters in total length with two 180 degree changes in direction. Between sprints, participants will have 10 seconds rest. After the first series of five sprints participants will be given a 2-minute rest interval. Then participants will perform another series of five sprints followed by another 2-minute rest interval. During each rest interval, Group A will utilize a palmar cooling device. Group B will utilize a placebo version of the palmar cooling device. All sprints will be timed. Heart rate recovery will be measured during all rest breaks, and a rating of perceived exertion will be measured at the beginning and end of each resting interval. Delayed onset muscle soreness will be assessed 48 hours post sprinting, utilizing a visual analog scale.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals 18-30 years of age

Exclusion Criteria:

* Participant self-reporting injury or illness that will prevent them from exercising at maximal capacity
* If participant has been told by their healthcare provider that they should avoid exercising at maximal capacity
* Has previously used the palmar cooling device

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2024-06-28 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Participants Sprinting times | 1 day

SECONDARY OUTCOMES:
Participants Heart Rate Recovery | 1 day
Participants Rating of Perceived exertion | 1 day
  Borg RPE Scale (6-20)
Participants Reported Delayed Onset Muscle Soreness | 2 days after the intervention
  Visual Analog Scale 1-10

CONTACTS AND LOCATIONS:
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: Undecided